CLINICAL TRIAL: NCT05355194
Title: Effects of Kinesiotaping With and Without Pelvic Tilts on Pain and Menstrual Distress in Females With Dysmenorrhea
Brief Title: Effects of Kinesiotaping With and Without Pelvic Tilts in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0505 Izza
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; Active stretching; Kinesiotape
MeSH Terms: conditions — Dysmenorrhea | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Kinesiotaping with pelvic tilts (Experimental): Kinesiotape will be applied to patients. In addition, patients will be instructed to perform pelvic tilts.
  Interventions: Other: Kinesiotape; Other: Pelvic Tilts
- Group B: Kinesiotaping without pelvic tilts (Active Comparator): Kinesiotape will be applied to patients.
  Interventions: Other: Kinesiotape

INTERVENTIONS:
Other: Kinesiotape — Patients will be instructed to inhale while taping the application. The tape will be applied in a vertical direction from just below the navel to the pubic region, another tape will be applied over the initial tape in the horizontal direction with minimal stretch. Another tape will be applied over the lumbosacral region making a V shape. The arms of V shall lie over the lumbar region while the base shall rest over the caudal region. Taping will be maintained for at least 48 hours.
  The interventions shall be applied for two consecutive menstrual cycles.
Other: Pelvic Tilts — Patients will be asked to lie in a supine position with legs bent and toes facing forward. Afterward, they will be instructed to pull their belly inwards while pushing pelvis towards the ceiling and keep hip muscles tightened. This position will be maintained for 5 seconds with 3 sets of 20 repetitions. Pelvic tilts must be performed throughout the menstrual cycle.
  Arms: Group A: Kinesiotaping with pelvic tilts

SUMMARY:
This study aims to determine the effects of kinesiotaping with & without pelvic tilts on pain & menstrual distress in females with dysmenorrhea. This study will be a randomized controlled trial to compare the effectiveness of kinesiotaping with and without pelvic tilts in subjects with primary dysmenorrhea.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial to compare the effectiveness of kinesiotaping with and without pelvic tilts in subjects with primary dysmenorrhea. Subjects with primary dysmenorrhea meeting the predetermined eligibility criteria will be divided into two groups using the random sequence generation method. Pre-intervention responses shall be taken during the first menstrual cycle using the Numeric Pain Rating Scale, WaLLID tool & Menstrual Distress Questionnaire.

Subjects in Group A shall be treated with kinesiotaping and pelvic tilts while subjects in Group B shall be treated with kinesiotaping only. Each subject will receive 02 treatment sessions during the second & third menstrual cycles. Post-intervention responses shall be recorded in the fourth menstrual cycle using the Numeric Pain Rating Scale, WaLLID tool & Menstrual Distress Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* Nulliparous
* Regular menstrual cycles
* Primary dysmenorrhea (diagnosed via WaLLID tool)

Exclusion Criteria:

* Allergic to kinesiotape
* Skin disorders
* Uterine fibroids
* Endometriosis
* Polycystic Ovarian Syndrome

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | up to 12 weeks
  The Numeric Pain Rating Scale (NPRS) is an outcome measure that is unidimensional measure of pain intensity in adults. It is segmented numeric version of Visual Analogue Scale (VAS) in which respondents select a whole number from 0-10 that best reflects the intensity of their pain.
WaLLID Scale: | up to 12 weeks
  Proposed in 2018 by Teherán et al., working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD; based on pain score and use of painkillers) is a combination of multiple scales, which has been developed with the goal of measuring the severity of dysmenorrhea and predicting the resultant activity limitation.
Menstrual Distress Questionnaire: | up to 12 weeks
  Menstrual Distress Questionnaire is a tool developed by Moss that measures the severity and symptoms associated with menstruation. Kim designed a revised version of Menstrual Distress Questionnaire to determine the type of discomfort during menstruation wit 35 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PhD*, Principal Investigator — Riphah International University
Locations (1):
- University of Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddish S. Dysmenorrhoea. Aust Fam Physician. 2006 Nov;35(11):842-4, 846-9. PMID 17099800
- [Background] Ju H, Jones M, Mishra G. The prevalence and risk factors of dysmenorrhea. Epidemiol Rev. 2014;36:104-13. doi: 10.1093/epirev/mxt009. Epub 2013 Nov 26. PMID 24284871
- [Background] Johnston L. Menstrual pain (dysmenorrhoea). Professional Nursing Today. 2014;18(1):13-4.
- [Background] Smith R, Kaunitz A. Primary dysmenorrhea in adult women: clinical features and diagnosis. Alphen aan den Rijn: Wolters Kluwer. 2015.
- [Background] Lundeberg T, Bondesson L, Lundstrom V. Relief of primary dysmenorrhea by transcutaneous electrical nerve stimulation. Acta Obstet Gynecol Scand. 1985;64(6):491-7. doi: 10.3109/00016348509156727. PMID 3904321
- [Background] Patel F, Dhupkar A. Effect of Kinesiotaping and Pelvic Tilts on Menstrual Symptom Questionnaire and Visual Analogue Scale in Primary Dysmenorrhoea in Females Aged 18-30 Years.
- [Background] Tomas-Rodriguez MI, Palazon-Bru A, Martinez-St John DRJ, Toledo-Marhuenda JV, Asensio-Garcia MDR, Gil-Guillen VF. Effectiveness of medical taping concept in primary dysmenorrhoea: a two-armed randomized trial. Sci Rep. 2015 Nov 13;5:16671. doi: 10.1038/srep16671. PMID 26564807
- [Background] Roozbahani RE, Najad RM. A comparison of the effect of stretching exercises and kinesio taping on the primary dysmenorrhea of high school girls. J Arak Uni Med Sci. 2015;18(97):1-8.
- [Background] Shahr-Jerdy S, Hosseini RS, Gh ME. Effects of stretching exercises on primary dysmenorrhea in adolescent girls. Biomedical Human Kinetics. 2012;4(1):127-32.
- [Background] Ahmadi Barati A, Farhadi L, Khalily M. Comparison of the Effect of Stretching Exercises and Combination of Massage-Stretching Exercises on Primary Dysmenorrhea of Female Students of Razi University of Kermanshah. Journal of Clinical Research in Paramedical Sciences. 2021;10(1).
- [Background] Arshad S, Qureshi MF, Deeba F, Sarshad S, Shiraz S, Farooq S, et al. To compare the effectiveness of taping technique and hydrotherapy in treatment of primary dysmenorrhea. Inter J Endor Health Sci Res. 2018;6(3):34-42.